CLINICAL TRIAL: NCT07122167
Title: Post-market Registry Study on the Safety and Efficacy of ZENFLEX Pro™ Peripheral Drug-eluting Stent System for Femoropopliteal Artery Lesion
Brief Title: Post-market Registry Study on the Safety and Efficacy of ZENFLEX Pro™ Peripheral Drug-eluting Stent System for Femoropopliteal Artery Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MDCECRO LLC (Network)
Collaborators: Zylox-Tonbridge Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE-02
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prospective, Multi-center, Single-arm. (Other)
  Interventions: Device: Peripheral Drug-eluting Stent System

INTERVENTIONS:
Device: Peripheral Drug-eluting Stent System — Drug-eluting stents (DES) are increasingly used in the treatment of PAD. These stentsare coated with antiproliferative drugs designed to provide mechanical support within the artery while releasing the drug gradually to reduce the risk of restenosis. Commonly used drugs include paclitaxel, sirolimus, and everolimus, which inhibit vascular smooth muscle cell proliferation, thereby reducing the likelihood of re-occlusion.

SUMMARY:
This is a prospective, multi-center, single-arm post-market study evaluating the safety and effectiveness of the ZENFLEX Pro™ Drug-eluting Stent in treating femoropopliteal artery stenosis or occlusion. A total of 153 subjects will be followed at 1, 6, and 12 months. The primary endpoint is primary patency at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 18 to 80 years, regardless of gender. (2) Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3, 4 or 5. (3) Subject (or legal guardian, if applicable) is willing and able to provide consent before to the performance of any study specific tests or procedures, has signed the consent form and agrees to attend all required follow-up visits.

Angiographic Inclusion Criteria:

Eligible subjects must meet all of the following angiographic criteria:

1. Stenotic, restenotic or occlusive lesion(s) located in the native superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) (i.e., within the P1 segment):

   1. Degree of stenosis ≥70% by visual angiographic assessment.
   2. Vessel diameter ≥4.0 mm and ≤6.5 mm.
   3. Total lesion length (or series of lesions) ≥ 10 mm and ≤ 140 mm (Note: Lesion segment(s) must be fully covered with one stent).
   4. Chronic total occlusion with a total lesion length of ≤120 mm.
2. Patent popliteal and infrapopliteal arteries, with single-vessel runoff or better, defined as at least one of the three vessels remaining patent (i.e., <50% stenosis) down to the ankle or foot.

Exclusion Criteria:

* Clinical exclusion criteria:

Subjects will be excluded from the study if any of the following conditions are present:

1. Pregnant or breastfeeding women, or women/men planning to conceive.
2. Subjects who have had or are planned for major amputation (at or above the ankle level).
3. Subjects known to be allergic or intolerant to materials used in the investigational device or treatment drugs, including nitinol, paclitaxel, aspirin, clopidogrel, heparin, rivaroxaban, contrast agents, etc.
4. Subjects with serum creatinine ≥2.5 mg/dL or currently undergoing dialysis.
5. Subjects with known, uncorrectable hemorrhagic disorders or severe coagulation dysfunction (prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≥2 times the upper limit of normal, or platelet count <80×10⁹/L).
6. Previously stented target lesion/vessel.
7. Target lesion/vessel previously treated with drug-coated balloon <12 months prior to enrollment.
8. Subjects with a life expectancy of less than 1 year.
9. Subjects who have received local or systemic thrombolysis treatment within 48 hours prior to enrollment.
10. Subjects diagnosed with major clinical diseases or unstable conditions within the past 3 months, such as severe heart failure, unstable angina, myocardial infarction, transient ischemic attack or stroke, severe neurological or psychiatric history, severe infections, gastrointestinal bleeding, or active disseminated intravascular coagulation.
11. Subjects currently participating in another clinical trial involving drugs or medical devices.
12. Subjects whom the investigator considers unsuitable for participation in the clinical trial.

Angiographic exclusion criteria:

1. Presence of aneurysm in the target vessel.
2. Heavily calcified lesions (Peripheral Arterial Calcium Scoring System [PACSS] grades 3-4).
3. The target lesion requires the use of plaque excision, laser, or other debulking devices that may damage the vessel intima.
4. The guidewire cannot pass through the target lesion, or percutaneous transluminal angioplasty (PTA) balloon cannot be used for pre-dilation.
5. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency at 12 months post-procedure | 12 Months
  Primary vessel patency is defined as a binary endpoint and will be determined to be a success when the duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) is ≤2.4 at the 12-month follow-up visit in the absence of clinically driven TLR or bypass of the target lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular, Chrzanów, Chrzanow, Poland

IPD SHARING:
Plan to Share IPD: Undecided